CLINICAL TRIAL: NCT05946694
Title: Comparison of UESCOPE VL 400, I-VIEW, Airtraq Videolaryngoscopes and Macintosh Laryngoscope for Tracheal Intubation in Simulated Out-of-Hospital Conditions: A Randomized Crossover Manikin Study
Brief Title: Comparison of UESCOPE VL 400, I-VIEW, Airtraq for Tracheal Intubation in Simulated Out-of-Hospital Conditions
Status: Completed | Type: Observational
Sponsor: Medical University of Lodz (Other)
Responsible Party: Principal Investigator, Tomasz Gaszynski, prof. dr hab., Medical University of Lodz
Other Study IDs: RNN/363/13/KB
Record Dates: First submitted 2023-06-16; First posted 2023-07-14 (Actual); Last update posted 2023-07-14 (Actual); Status verified 2023-07

CONDITIONS: Training Group, Sensitivity
Keywords: laryngoscopy; endotracheal intubation; manikin study; videolaryngoscopes
MeSH Terms: conditions — Hypersensitivity | interventions — Intubation; Manikins

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- students: 30 students of the third year of Emergency Medicine, full-time first-degree program at the Medical University of Lodz, Poland, were enrolled in the study.
  Interventions: Other: intubation in manikin

INTERVENTIONS:
Other: intubation in manikin — Evaluation of 3 videolaryngoscopes under simulated out-of-hospital conditions by people without clinical experience on a manikin model

SUMMARY:
In the study, three videolaryngoscopes: UESCOPE VL 400 (Zhejiang UE Medical Corp. Zhejiang, China), I-View™ VL (Intersurgical Ltd, Wokingham, Berkshire, UK), Airtraq sp® (Prodol Meditec S.A, Vizcaya, Spain) were compared with the most widely used, classic Macintosh laryngoscope (HEINE Optotechnik GmbH & Co. KG, Gilch-ing, Germany) under simulated out-of-hospital conditions by people without clinical experience on a manikin model (Laerdal Airway Management Trainer Stavanger Norway manikin of universal difficulty), while using an endotracheal tube without and with a stylet. Simulated out-of-hospital conditions were created by placing the manikin at floor level. A random selection of 30 students of the third year of Emergency Medicine, full-time first-degree program at the Medical University of Lodz, Poland, were enrolled in the study. The following were assessed: intubation efficiency, time to ventilation (primary endpoints); intubation effort, intubator comfort, tooth damage and visibility of the glottis according to the Cormack-Lehane scale (secondary endpoints).

DETAILED DESCRIPTION:
Pre-study preparation All participants attended a 30-minute lecture on laryngoscope construction, principles of usage, anatomical structure of the airways, and intubation techniques. Following the lecture, the instructor demonstrated proper intubation using each of the four laryngoscopes that were being tested. Next, the students participated in a supervised workshop where they had the opportunity to intubate a mannequin placed on an operating table at an optimal height using each of the tested laryngoscopes with and without a stylet. One month later, 30 students participated in the actual study.

Simulation model To create simulated out-of-hospital conditions, a certified airway training manikin (Laerdal Airway Management Trainer Stavanger Norway of universal difficulty) was placed in a neutral position at floor level.

The trial tested three unchanneled videolaryngoscopes: UESCOPE VL 400 (Zhejiang UE Medical Corp. Zhejiang, China), I-View™ VL (Intersurgical Ltd, Wokingham, Berkshire, UK), Airtraq sp ® (Prodol Meditec S.A, Vizcaya, Spain), and a Macintosh laryngoscope (HEINE Optotechnik GmbH & Co. KG, Gilch-ing, Germany) (see Fig. 1).

Each participant performed eight intubations on the manikin using all four devices. The intubation order was randomized using a blocked randomization strategy generated by the Randomizer Program (randomizer.org). A sealed opaque envelope was used to determine the order in which the laryngoscopes were used, and whether the tube was with or without a stylet.

After each intubation, there was a minimum 10-minute pause before the next one. The subject then proceeded to the next intubation with the randomly selected laryngoscope, with the tube and stylet as determined by the sealed envelope.

All intubations were performed using a polyvinyl chloride cuffed endotracheal tube (Covidien LLC, Hampshire Street, Mansfield, USA; internal diameter 7.0 mm) and an endotracheal stylet (Sumi® from sp. z o.o., 35 Drobiarska Street, 05-070 Sulejówek, Poland), when used. The endotracheal tubes and stylets were coated with a standard lubricant for simulators. All data were pseudonymized for each simulation.

The time was measured by the same investigator (P.R.) using a stopwatch for all TI attempts. The timing measurement started when the participant picked up the laryngoscope and ended when initial ventilation was achieved using a resuscitation bag after the placement and sealing of the endotracheal tube. Successful TI was confirmed by observing the breathing movements of the manikin lungs. An unsuccessful attempt was defined by the absence of respiratory movements of the dummy or an intubation time of more than 60 seconds. This criterion was adopted because the study aimed to assess the suitability of the devices for individuals without clinical experience in intubation. Participants without sufficient skills or a good view of the glottis could prolong intubations without knowing how to solve the problem. In a real clinical scenario, such prolongation of intubation attempts beyond 60 seconds could result in irreversible brain damage in the victim, especially considering the necessary time for the emergency medical team to arrive.

Participants rated the level of effort required to perform TI using the modified Borg scale (0 - no effort, 10 - maximum effort) and graded their comfort during the procedure as "full comfort, satisfactory comfort, moderate comfort, unsatisfactory comfort, and no comfort."

ELIGIBILITY:
Inclusion Criteria:

* attaneding students

Exclusion Criteria:

* lack of conscent to participate

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: intubation effort, intubator comfort, tooth damage and visibility of the glottis according to the Cormack-Lehane scale
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-01 (Actual); Study Completion 2023-02-01 (Actual)

PRIMARY OUTCOMES:
time to ventilation | during the procedure
  time from grabbing the laryngoscope to confirmed intubation measured in sec
intubation efficacy | during the procedure
  endotracheal intubation confirmed by ventilation of manikin's lungs, measured yes/no

SECONDARY OUTCOMES:
intubation effort | during the procedure
  how many intubations are required to success, measured in number of attempts
intubator comfort, | during the procedure
  operator's experience measured with Borg scale
tooth damage | during the procedure
  tooth damage recorded by manikin sensors, measured yes/no
visibility of the glottis according to the Cormack-Lehane scale | during the procedure
  visibility of glottis in Cormack-Lehane score assessed by operators, measured using Cormack-Lehane scale

CONTACTS AND LOCATIONS:
Overall Officials: Tomasz Gaszynski, Prof, Principal Investigator — Medical University of Lodz, Poland
Locations (1):
- Medical University of Lodz, Poland, Lodz, Poland

IPD SHARING:
Plan to Share IPD: Undecided